CLINICAL TRIAL: NCT04974606
Title: Effect of Coffeeberry on Mood, Motivation and Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-1605
Record Dates: First submitted 2021-07-09; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Fatigue, Mental; Alertness; Mood; Motivation; Cognitive Performance
Keywords: alertness; mental fatigue; coffeeberry; coffee fruit
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Coffeeberry 100 mg beverage (Experimental): Appearance-matched to the other beverages
  Interventions: Dietary Supplement: Cherry-flavored still beverage
- Coffeeberry 300 mg beverage (Experimental): Appearance-matched to the other beverages
  Interventions: Dietary Supplement: Cherry-flavored still beverage
- Placebo beverage (Placebo Comparator): Appearance-matched to the other beverages
  Interventions: Other: Placebo cherry-flavored still beverage
- Caffeine 75 mg beverage (Active Comparator): Appearance-matched to the other beverages
  Interventions: Dietary Supplement: Cherry-flavored still beverage

INTERVENTIONS:
Dietary Supplement: Cherry-flavored still beverage — 10 oz bottle
  Arms: Caffeine 75 mg beverage; Coffeeberry 100 mg beverage; Coffeeberry 300 mg beverage
Other: Placebo cherry-flavored still beverage — 10 oz bottle
  Arms: Placebo beverage

SUMMARY:
The primary purpose is to test the short-term effects of the acute consumption of two novel beverages made from coffeeberries, the fruit of the coffee plant (Coffea arabica) benchmarked against caffeine on several aspects of cognitive performance.

Preliminary studies suggest that flavanols and chlorogenic acids can enhance cognitive performance. It is unknown if drinks formulated with flavanols and chlorogenic acids (without high sugar or caffeine) improve cognition or mood to a similar extent as caffeine. Coffeeberry beverage comparisons will be made to a flavored positive control beverage containing caffeine and a flavored placebo beverage.

ELIGIBILITY:
Inclusion Criteria:

* Are older than 17 and under 50 years of age
* Self-report of good health

Exclusion Criteria:

* Using any prescription medication including birth control
* Report hypersensitivity to caffeine
* Have visual impairment that cannot be corrected with glasses or contact lenses
* Report any food allergies
* Self-reported excessive leisure time physical activity (> 7 strenuous bouts per week)
* the presence of current gastrointestinal, sleep, or psychiatric disorder,
* Report pregnancy/lactation, illegal drug use, smoker
* failure to demonstrate adequate minimal performance on lab, computer-based cognitive tasks.
* Participation in another clinical trial within past 30 days

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2016-12-16 (Actual); Study Completion 2016-12-16 (Actual)

PRIMARY OUTCOMES:
Cognition score | Change from baseline to 60 and 120 min post-consumption. Higher test scores are better.
  Objective Cognitive Demand Battery (CDB) using Computerised Mental Performance Assessment framework tasks (COMPASS) for word and picture presentation and recall, serial 3 and 7 subtraction, Rapid Visual Information Processing (RVIP).
Fatigue score | Change from baseline to 60 and 120 min post-consumption. Lower fatigue score is better.
  Subjective Visual Analog Scale (VAS) rating from 1-100 mm from not at all to extremely, during Cognitive Demand Battery (CDB) using Computerised Mental Performance Assessment framework tasks (COMPASS)
Alertness score | Change from baseline to 60 and 120 min post-consumption. Higher alertness score is better.
  Subjective Bond-Lader Visual Analog Scale (VAS) rating from 1-100 mm representing the full range of each dimension from not at all to extremely, during Cognitive Demand Battery (CDB) Visual Analog Scale (VAS) rating from 1-100 mm during Cognitive Demand Battery(CDB) within Computerised Mental Performance Assessment framework tasks (COMPASS)
Calmness score | Change from baseline to 60 and 120 min post-consumption. Higher calmness score is better.
  Subjective Bond-Lader Visual Analog Scale (VAS) rating from 1-100 representing the full range of each dimension from not at all to extremely, during Cognitive Demand Battery (CDB)during Cognitive Demand Battery (CDB) Visual Analog Scale (VAS) rating from 1-100 mm during Cognitive Demand Battery(CDB) within Computerised Mental Performance Assessment framework tasks (COMPASS)
Contentedness score | Change from baseline to 60 and 120 min post-consumption. Higher contentedness score is better.
  Subjective Bond-Lader Visual Analog Scale (VAS) rating from 1-100 mm representing the full range of each dimension from not at all to extremely, during Cognitive Demand Battery (CDB)during Cognitive Demand Battery (CDB) Visual Analog Scale (VAS) rating from 1-100 mm during Cognitive Demand Battery(CDB) within Computerised Mental Performance Assessment framework tasks (COMPASS)
Motivation score | Change from baseline to 60 and 120 min post-consumption. Higher motivation score is better.
  Subjective Visual Analog Scale (VAS) rating from 1-100 mm from not at all to extremely, during Cognitive Demand Battery (CDB) within Computerised Mental Performance Assessment framework tasks (COMPASS)
Energy score | Change from baseline to 60 and 120 min post-consumption. Stronger feelings of mental and physical energy are better.
  Subjective mental and physical state energy and fatigues scales (EFS-State Scale). Composite scores range from 0 to 300 mm, from feelings of no energy to strongest feelings of energy during Cognitive Demand Battery (CDB) using Computerised Mental Performance Assessment framework tasks (COMPASS)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J O'Connor, Principal Investigator — University of Georgia, Athens
Locations (1):
- Exercise Psychology Laboratory University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No